CLINICAL TRIAL: NCT02181023
Title: Acute Effect of Aclidinium on Hyperinflation and Lung Volume Distribution in Severe COPD Patients
Brief Title: Acute Effect of Aclidinium on Hyperinflation and Ventilation Inhomogeneity in Severe COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Pierachille Santus, Head of Pulmonary Rehabilitation Unit, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 960CEC
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Hyperinflation; Aclidinium; Glycopyrronium; Volume distribution; Anticholinergic; Pharmacokinetics; Single Breath Nitrogen Test; Phase III
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aclidinium - Glycopyrronium (Experimental): Patients will assume Aclidinium Bromide 322 dry powder by Genuair inhaler and Glycopyrronium 44 dry powder inhaler by Breezehaler inhaler (placebo) after 72 hours from inhalatory therapy washout (only short acting bronchodilators permitted). Then, after 72 hours of inhalatory drugs washout (only short acting bronchodilators permitted), they will receive Glycopyrronium Bromide 322 mcg via Breezehaler inhaler and Aclidinium Bromide 322 dry powder by Genuair inhaler (placebo).
  Interventions: Drug: Aclidinium Bromide; Drug: Glycopyrronium Bromide
- Glycopyrronium - Aclidinium (Experimental): Patients will assume Glycopyrronium Bromide 44 mcg dry powder by Breezehaler inhaler and Aclidinium Bromide 322 dry powder by Genuair inhaler (placebo) after 72 hours of inhalatory therapy washout (only short acting bronchodilators permitted). Then, after 72 hours of inhalatory drugs washout (only short acting bronchodilators permitted) they will receive Aclidinium Bromide 322 mcg via Genuair inhaler and Glycopyrronium Bromide 44 mcg dry powder by Breezehaler inhaler (placebo).
  Interventions: Drug: Aclidinium Bromide; Drug: Glycopyrronium Bromide

INTERVENTIONS:
Drug: Aclidinium Bromide — Aclidinium Bromide 322 mcg inhalation powder via Genuair inhaler (Eklira) Product by Almirall, S.A. Ronda General Mitre, 151. ES-08022 Barcelona, Spain
  Other Names: Eklira Genuair (UK); Tudorza Pressair (US); Bretaris Genuair (EU)
Drug: Glycopyrronium Bromide — Glycopyrronium Bromide 44 mcg dry powder (capsules) inhaled via Breezehaler inhaler, Seebri - product by Novartis Europharm Limited - Wimblehurst Road, Horsham, West Sussex, RH12 5AB; United Kingdom
  Other Names: Seebri Breezhaler

SUMMARY:
* Chronic Obstructive Pulmonary Disease (COPD) is characterized by lung hyperinflation and flow limitation. These physiopathological modifications are secondary to loss of elastic recoil and bronchial obstruction due to emphysema.
* The cornerstone of COPD treatment is represented by inhaled beta-2 agonists and anticholinergics. The molecules of the latter classes can be characterized by short lasting action (few hours), long acting action (12 hours) or ultra long acting duration of action (24 hours).
* For years the only anticholinergic (or antimuscarinic) drug other than those used by aerosol, was Tiotropium Bromide. Recently two new antimuscarinic agents have been launched on the market: glycopyrronium bromide (once daily) and aclidinium (twice daily).
* The Single Breath Nitrogen Test is capable of identifying the pulmonary closing volume. The part of the curve that reflects lung ventilation inhomogeneity is the slope of phase III
* For COPD patients, the most important characteristic for an inhalatory drug is a prompt action in order to give a quick relief from respiratory symptoms, in particular dyspnoea.
* The objective of this study is to study the acute action of glycopyrronium and aclidinium in terms of reduction of hyperinflation, pulmonary specific resistances, lung volume distribution and dyspnoea at rest in severe COPD patients.
* To our knowledge no study has explored these aspects before.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a disease characterized by progressive and evolutionary physiopathological changes that are responsible for the developing of respiratory symptoms, disability, poor quality of life and morbidity. These changes are secondary to parenchymal disruption and chronic bronchiolar inflammation in major part due to cigarette smoke.

Lung architectural derangement and loss of elastic recoil secondary to emphysema together with decreased internal bronchiolar lumen due to mucosal chronic inflammation are responsible for bronchial obstruction, flow limitation and lung hyperinflation. All these features bring to exertional dyspnoea, chronic cough and sputum and so decreased activeness in daily life activities.

The Single Breath Nitrogen Washout Test (SBN2) is one of the test that more adequately can catch the modifications of small airways and their premature collapse called closing volume (CV). Together with CV the test reflects pulmonary ventilation inhomogeneity through the slope of the so called phase III (a plateau line of nitrogen concentration that is steeper the bigger the ventilation inhomogeneity). In literature the effects of COPD inhalatory treatments on this modifications and on hyperinflation were until today poorly analysed. Recently some new anticholinergic molecules were developed, in particular Aclidinium Bromide and Glycopyrronium Bromide, and there is no trace of such evaluation in medical literature with those new inhalatory drugs.

The study of the acute effects of these drugs on lung mechanics are mandatory because the quicker the effects, the faster the patient's dyspnoea relief.

The study will comprise a first enrollment visit and then the suitable subjects will undergo a pharmacological washout of 72 hours from any inhalatory drug except from Salbutamol.

Then the patients will be randomised to be given Glycopyrronium Bromide 44 mcg (and matched Aclidinium Bromide 322 mcg placebo) or Aclidinium Bromide 322 mcg (and matched Glycopyrronium Bromide 44 mcg placebo) (Day 1) with a double dummy scheme.

At day 1 the pre-dose (baseline) evaluation consists of:

* body plethysmography (with residual volume and specific resistances evaluation),
* arterial blood gas analysis (partial pressure of oxygen and carbon dioxide evaluation),
* SBN2
* Visual Analogic Scale for Dyspnoea (VAS scale) evaluation
* Diffusion Lung Capacity for Carbon Monoxide with Single Breath method (DLCO). These tests will be repeated after 5, 15, 30, 60 and 180 minutes after study drug inhalation. DLCO and arterial blood gas analysis will be performed only at baseline and after 180 minutes after study drug inhalation.

After day 1 all the patients will undergo another period of inhalatory therapy washout of 72 hours (only rescue Salbutamol spray permitted).

After the second pharmacological washout the patients will undergo the crossing over. The ones who were given Aclidinium Bromide will assume Glycopyrronium Bromide and vice versa (Day 2) always in double dummy conditions.

At Day 2 all the patients will undergo the same evaluation as in day 1. At day 1 and day 2 the study drugs with the two different devices (active drug + placebo) will be given to the patients by medical personnel not involved in the performing of any of the tests of day 1 and 2, in order to maintain the double blind conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* COPD patients with age raging from 50 to 85 years old
* Patients with at least a history of COPD of one year
* COPD patients clinically stable in the last three months
* COPD subjects with Forced Expiratory Volume at one second (FEV1)<50% of predicted value
* COPD subjects with Residual Volume (RV) >125% predicted value
* FEV1/Forced Vital Capacity (FVC) <88% (males) or <89% (females) of Low Levels of Normality (LLN)
* COPD former or active smokers with at least a smoking history of 20 pack year

Exclusion Criteria:

* Acute Bronchial Exacerbation at recruitment
* Fertile women with age between 18 and 50 years old or with active period
* Pregnancy
* Subjects enrolled in other clinical trials or that have taken part in one of them in the month preceding the enrollment.
* FEV1/FVC more than 70% of predicted value in basal conditions
* FEV1 more than 70% of predicted value in basal conditions
* Known deficit of alpha 1 antitrypsin
* Subjects that underwent a Lung Volume Reduction Surgery (LVRS)
* Subjects with known positivity to Human Immunodeficiency Virus (HIV)
* Misuse of alcool or drugs
* Lack of compliance in performing respiratory tests
* Subjects not capable to follow the study prescriptions because of psychic disorders or language problems.
* Long Term Oxygen Therapy with flows > 6 litres per minute (l/min) at rest

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Residual Volume Variation from baseline | At baseline, 5, 15, 30, 60 and 180 minutes after study drug administration
  Residual Volume is obtained by performing body plethysmography before study drug inhalation (baseline), and again 5, 15, 30,60 and 180 minutes after inhalation of study drug. The same subject will undergo the same evaluation in the second part of the study, after the crossing over
Functional Residual Capacity variation from baseline | At baseline, 5, 15, 30, 60 and 180 minutes after study drug administration
  Functional Residual Capacity (plethysmographic Intra Thoracic Gas Volume - ITGV) is obtained by performing body plethysmography before study drug inhalation (baseline), and again 5, 15, 30,60 and 180 minutes after inhalation of study drug. The same subject will undergo the same evaluation in the second part of the study, after the crossing over

SECONDARY OUTCOMES:
Phase III slope variation from baseline | At baseline, 5, 15, 30, 60 and 180 minutes after study drug administration
  Phase III slope is measured from the Single Breath Nitrogen Washout curve. It is measured at baseline (before study drug administration, and after 5, 15, 30, 60 and 180 minutes after study drug administration. The same patient will perform the same evaluation after drug crossing over
Visual Analogical Scale (VAS) for Dyspnoea at rest variation from baseline | At baseline, 5, 15, 30, 60 and 180 minutes after study drug administration
  Visual Analogical Scale (VAS) for Dyspnoea is obtained by asking the patients to evaluate the intensity of dyspnoea sensation at rest putting a sign in a scale that ranges from 0 to 10, being 10 the maximum dyspnoea discomfort and 0 the absence of dyspnoea sensation. The VAS scale will be performed before study drug inhalation (baseline), and again 5, 15, 30,60 and 180 minutes after inhalation of study drug. The same subject will undergo the same evaluation in the second part of the study, after the crossing over.
Oxygen and Carbon Dioxide variation from baseline | At baseline and 180 minutes after inhalation of study drug
  Partial Pressure of Oxygen (PaO2) and Partial Pressure of Carbon Dioxide (PaCO2) are obtained from arterial blood gas analysis before study drug inhalation and 180 minutes after drug inhalation. Patients will undergo the same evaluation after drug crossing over

OTHER OUTCOMES:
Specific AirWay Resistances (sRAW) variation from baseline | At baseline, 5, 15, 30, 60 and 180 minutes after study drug administration
  Specific AirWay Resistances (sRAW) are calculated from body plethysmography before study drug inhalation (baseline), and again 5, 15, 30,60 and 180 minutes after inhalation of study drug. The same subject will undergo the same evaluation in the second part of the study, after the crossing over

CONTACTS AND LOCATIONS:
Overall Officials: Pierachille Santus, MD, PhD, Study Director — Università degli Studi di Milano-Pneumologia Riabilitativa-Fondazione Salvatore Maugeri-MILANO
Locations (1):
- Fondazione Salvatore Maugeri, Milan, Milan, Italy

REFERENCES:
- [Derived] Santus P, Radovanovic D, Di Marco F, Raccanelli R, Valenti V, Centanni S. Faster reduction in hyperinflation and improvement in lung ventilation inhomogeneity promoted by aclidinium compared to glycopyrronium in severe stable COPD patients. A randomized crossover study. Pulm Pharmacol Ther. 2015 Dec;35:42-9. doi: 10.1016/j.pupt.2015.11.001. Epub 2015 Nov 6. PMID 26549785